CLINICAL TRIAL: NCT04034251
Title: A Phase II Study of Intraperitoneal and Intravenous Paclitaxel Chemotherapy With Oral Capecitabine for Gastric Adenocarcinoma With Peritoneal Carcinomatosis
Brief Title: Intraperitoneal and Intravenous Paclitaxel Chemotherapy With Oral Capecitabine for Gastric Adenocarcinoma With Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Blakely, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190129; 19-C-0129
Record Dates: First submitted 2019-07-25; First posted 2019-07-26 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer; Esophagogastric Junction; Peritoneal Carcinomatosis
Keywords: Gastroesophageal Junction (Siewert III) Adenocarcinoma; Intravenous Chemotherapy; Progression Free Survival; Peritoneal Metastasis; Intraperitoneal Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms; Adenocarcinoma | interventions — Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily (Experimental): Intraperitoneal (IP) and intravenous (IV) paclitaxel administration with concomitant oral capecitabine
  Interventions: Drug: Paclitaxel; Drug: Capecitabine; Device: BardPort Titanium Implanted Port with Peritoneal Catheter
- Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily (Experimental): Intraperitoneal (IP) and intravenous (IV) paclitaxel administration with concomitant oral capecitabine
  Interventions: Drug: Paclitaxel; Drug: Capecitabine; Device: BardPort Titanium Implanted Port with Peritoneal Catheter
- Paclitaxel Intraperitoneal & Intravenous Every 3 Weeks & Capecitabine Twice Daily (Experimental): Intraperitoneal (IP) and intravenous (IV) paclitaxel administration with concomitant oral capecitabine
  Interventions: Drug: Paclitaxel; Drug: Capecitabine; Device: BardPort Titanium Implanted Port with Peritoneal Catheter

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel (intraperitoneal (IP) and intravenous (IV), Day 1 of each 3-week cycle: Paclitaxel IP - Intraperitoneal paclitaxel (60 mg/m^2) will be diluted in 500 mL of 0.9% normal saline (NS), to be infused as rapidly as tolerated once per 3-week cycle on Day 1. Paclitaxel IV - Intravenous paclitaxel (80 mg/m^2) will be administered concomitantly over 3 hours, diluted in 100 to 250 ml of 0.9% NS once per 3-week cycle on Day 1.
  Other Names: Taxol
Drug: Capecitabine — Day 1-15 of each 3-week cycle: oral capecitabine (825 mg/m^2) to be taken twice a day starting the evening of Day 1 of each cycle until the morning of Day 15, followed by a 7-day rest period during each 3-week cycle.
  Other Names: Xeloda
Device: BardPort Titanium Implanted Port with Peritoneal Catheter — After peritoneal chemo infusion port is placed (Days 1-3, as dictated by clinical status), patients will begin intraperitoneal paclitaxel and intravenous paclitaxel (Day 1) followed by oral capecitabine on the evening of Day 1 to the morning of Day 15.

SUMMARY:
Background:

Three-fourths of people diagnosed with gastric cancer will die from it. Researchers want to see if giving cancer drugs in a new way can help people live longer and delay the time it takes for the cancer to grow.

Objective:

To find a better way to treat advanced stomach cancer.

Eligibility:

People ages 18 and older with stomach cancer that has spread throughout their belly.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, urine, and heart tests

Scans

Cancer sample: If they do not have one, they will have a biopsy.

Tests of performance of normal activities

Dietary assessment

Participants will have a laparoscopy. Small cuts are made into their abdomen. A thin camera with a light is inserted. Small instruments are used to take biopsies. This will be repeated during the study to monitor the cancer. During the first laparoscopy, a port with a catheter attached will be put into the abdomen.

Participants may also have an endoscopy: A thin tube with a camera is inserted through the mouth and into the stomach. The tube collects samples to monitor the cancer.

Participants will get paclitaxel every 3 weeks through the abdominal port and through a small plastic tube in an arm vein. They will also take capecitabine by mouth twice daily for the first 15 days of a 21-day cycle.

After participants finish 3 cycles, they will have scans to see how they are doing. They may get another course of therapy.

Participants will have visits every 3 weeks during treatment. Then they will have follow-up visits for 5 years. Then they will keep in touch with researchers for the rest of their life.

DETAILED DESCRIPTION:
Background:

* An estimated 28,000 cases of gastric adenocarcinoma are diagnosed annually in the United States (U.S.)
* Peritoneal metastasis is a common finding at diagnosis, making curative surgical resection possible in an estimated 25% of patients.
* Systemic chemotherapy is the recommended treatment for patients with metastatic gastric cancer to the peritoneal cavity, however selective use of cytoreductive surgery and intraperitoneal chemotherapy has been associated with improved overall survival.
* Multiple chemotherapeutic agents and delivery systems have been described for intraperitoneal therapy, but no standard regimen exists.

Objective:

-Determine the intraperitoneal progression free survival (iPFS) in patients with peritoneal metastases from gastric cancer after repeated intraperitoneal chemotherapeutic infusion (IPC) and systemic paclitaxel administration with concomitant capecitabine therapy.

Eligibility:

* Histologically confirmed adenocarcinoma of the stomach.
* Radiographic evidence of peritoneal carcinomatosis and/or sub-radiographic evidence of peritoneal carcinomatosis found at staging laparoscopy.
* Medically fit for systemic chemotherapy and intraperitoneal chemotherapy.
* Men and women age greater than or equal to 18 years.

Design:

* Phase II, nonrandomized, open label study.
* Patients will enroll in two cohorts: those with prior systemic chemotherapy and those who are treatment naive.
* Patients undergo staging laparoscopy and placement of peritoneal access port.
* Intraperitoneal paclitaxel (60 mg/m^2 weekly), intravenous paclitaxel (80 mg/m^2 weekly), and capecitabine (825 mg/m^2 twice daily for 14 days of each cycle) for 12 weeks.
* Treatment response will be assessed with imaging and laparoscopy.
* It is expected that 16-20 patients per year for total 4 years will be enrolled. The accrual ceiling is set at 74 patients.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologically or cytologically confirmed gastric adenocarcinoma, including Siewert III gastroesophageal junction adenocarcinoma, confirmed by the National Cancer Institute (NCI) Laboratory of Pathology, and have provided a block or unstained slides of primary or

   metastatic tumor tissue or newly obtained fresh biopsy of a tumor lesion in case archival tissue sample is not available.
2. Patients may be treatment naive or have received systemic chemotherapy prior to enrollment:

   * Trastuzumab allowed as prior treatment for human epidermal growth factor receptor 2 (HER2)/neu over-expressing cancers as clinically indicated.
   * Last dose of chemotherapy at least 2 weeks prior to enrollment with recovery to Grade 1 from chemotherapy-related toxicities.
3. Radiographic evidence of peritoneal carcinomatosis and/or sub-radiographic evidence of peritoneal carcinomatosis found at staging laparoscopy.
4. Age >=18 years. Children under the age of 18 will not participate in this study as gastric cancer is rare in this population.
5. Eastern Cooperative Oncology Group (ECOG) performance status <=1
6. Patients must have normal organ and marrow function as defined below:

   hemoglobin >=8.0 g/dL

   absolute neutrophil count >=1,000/mcL

   platelets >=100,000/mcL

   total bilirubin <=1.5 X institutional upper limit of normal

   Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) <=2.5 X institutional upper limit of normal

   creatinine <1.5 mg/dl

   OR

   creatinine clearance >=60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
7. Physiologically able to undergo laparoscopy and systemic chemotherapy.
8. Ability of subject to understand and the willingness to sign a written informed consent document.
9. Previous exploratory laparotomy or laparoscopy with tissue biopsy or peritoneal lavage is permitted.
10. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
11. Patients must be co-enrolled in protocol 13C0176 (NCT01915225) and 17C0044 (NCT03027427) for sample collection.
12. Human immunodeficiency virus (HIV)-positive patients may be considered for this study only after consultation with a National Institute of Allergy and Infectious Diseases (NIAID) physician.

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents.
2. Previous cytoreductive surgery or intraperitoneal chemotherapy.
3. Disseminated extra-peritoneal or solid organ metastases:

   * Excludes greater omentum and ovarian metastases.
   * Radiographic signs or clinical symptoms consistent with malignant bowel obstruction.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Paclitaxel or Capecitabine or other agents used in study.
5. Previous treatment with paclitaxel or nab-paclitaxel resulting in progression of disease.
6. Existing peripheral neuropathy, Grade 3 or greater.
7. Past medical history of dihydropyrimidine dehydrogenase deficiency.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant women are excluded because paclitaxel and capecitabine can cause fetal harm when administered to pregnant women. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel and capecitabine, breastfeeding should be discontinued if the mother is treated with paclitaxel and capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0129.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily: Intraperitoneal and intravenous paclitaxel administration with concomitant oral capecitabine.
  Intraperitoneal Paclitaxel (20 mg/m^2) every 3 weeks (Q3WK), intravenous Paclitaxel (80 mg/m^2) Q3WK, Capecitabine (825mg/m^2 twice daily (BID) x 14 days of each cycle).
  Cohort A: Participants with confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction (Siewert III) adenocarcinoma who have received prior systemic chemotherapy.
- Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily: Intraperitoneal and intravenous paclitaxel administration with concomitant oral capecitabine.
  Intraperitoneal Paclitaxel (60 mg/m^2) every 3 weeks (Q3WK), intravenous Paclitaxel (80 mg/m^2) Q3WK, Capecitabine (825mg/m^2 twice daily (BID) x 14 days of each cycle).
  Cohort A: Participants with confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction (Siewert III) adenocarcinoma who have received prior systemic chemotherapy.
- Paclitaxel Intraperitoneal & Intravenous Every 3 Weeks & Capecitabine Twice Daily: Intraperitoneal and intravenous paclitaxel administration with concomitant oral capecitabine.
  Cohort B: Participants with confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction (Siewert III) adenocarcinoma who have received prior systemic chemotherapy.
Period: Overall Study
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal & Intravenous Every 3 Weeks & Capecitabine Twice Daily
Started | 5 | 7 | 0 (No participants were enrolled on Cohort B.)
Completed | 4 | 7 | 0
Not Completed | 1 | 0 | 0
Not completed — Screen failure due to development of solid organ mets in lung; no longer met eligibility criteria. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Collected baseline data are reported for one participant in the first group who was later deemed ineligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.28 (9.79) | 50.39 (7.98) | 49.51 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in Participants With Peritoneal Metastases From Gastric Cancer After Repeated Intraperitoneal Chemotherapeutic Infusion (IPC) and Systemic Paclitaxel Administration With Concomitant Capecitabine Therapy
Description: PFS is the amount of time a participant survives without progression of disease after treatment with peritoneal metastases from gastric cancer after repeated intraperitoneal chemotherapeutic infusion (IPC) and systemic paclitaxel administration with concomitant capecitabine therapy. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as an increase in peritoneal cancer index (PCI) score of greater than 4 points from baseline PCI, new ascites requiring repeat (more than 1) therapeutic paracentesis, malignant bowel obstruction, new intraperitoneal nodules or masses concerning for peritoneal metastasis, and decline in performance status not attributable to other medical causes.
Time Frame: From the first treatment to progression of disease, up to 2 years and 1 month
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Median (Full Range); unit: Months
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Months | 4.2 [1.5 to NA] — NA = It is not estimable because there are insufficient events after the median is identified for the upper bound of the confidence interval to be computed. This is mostly a situation when there are very few participants, or virtually all events take place before the median time. | 13.3 [1.5 to 13.3]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is the median amount of time a participant survives after treatment.
Time Frame: From first treatment until death, an average of 1.5 years
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Months | 10.6 [4.7 to 12.5] | 14.7 [4.0 to 17.7]

3. Secondary Outcome: Number of Grades 3-5 Serious and/or Non-serious Adverse Events Related to the Research Interventions
Description: Serious and/or non-serious adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death.
Time Frame: Date treatment consent signed to date off study, 18 months and 8 days; and 25 months and 10 days for the first and second group, respectively.
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Number; unit: adverse events
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
adverse events
  Serious Adverse Events Grade 3 | 0 | 1
  Serious Adverse Events Grade 4 | 0 | 0
  Serious Adverse Events Grade 5 | 0 | 0
  Non-Serious Adverse Events Grade 3 | 8 | 7
  Non-Serious Adverse Events Grade 4 | 0 | 1

4. Secondary Outcome: Intra-peritoneal Progression Free Survival (iPFS) Reported With an 80% Confidence Interval
Description: iPFS is the median amount of time a participant survives without intra-peritoneal disease progression reported with an 80% confidence interval. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as an increase in peritoneal cancer index (PCI) score of greater than 4 points from baseline PCI. New ascites requiring repeat (more than 1) therapeutic paracentesis, malignant bowel obstruction, new intraperitoneal nodules or masses concerning for peritoneal metastasis, and decline in performance status not attributable to other medical causes.
Time Frame: From the first treatment to progression of disease, up to 2 years and 1 month
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Months | 4.2 [1.4 to NA] — NA=It is not estimable because there are insufficient events after the median is identified for the upper bound of the confidence interval to be computed. This is mostly a situation when there are very few participants, or virtually all events take place before the median time. | 13.3 [2.1 to 13.3]

5. Secondary Outcome: Intra-peritoneal Progression Free Survival (iPFS) Reported With an 95% Confidence Interval
Description: Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as an increase in peritoneal cancer index (PCI) score of greater than 4 points from baseline PCI. New ascites requiring repeat (more than 1) therapeutic paracentesis, malignant bowel obstruction, new intraperitoneal nodules or masses concerning for peritoneal metastasis, and decline in performance status not attributable to other medical causes.
Time Frame: From the first treatment to progression of disease, up to 2 years and 1 month
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Months | 4.2 [1.4 to NA] — NA = It is not estimable because there are insufficient events after the median is identified for the upper bound of the confidence interval to be computed. This is mostly a situation when there are very few participants, or virtually all events take place before the median time. | 13.3 [1.5 to 13.3]

6. Secondary Outcome: Frequency of Objective Histopathologic Response to Therapy
Description: Participants metastatic tumors are biopsied at the end of a course of therapy and graded according to standard pathologic technique.
Time Frame: At end of each course (3 treatment cycles; 9 weeks)
Population: No data was collected. The pathologists were not able to provide an objective measure for this information due to technical reasons.
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Distant Extra-peritoneal Disease-free Survival
Description: dDFS was determined based on identification of only distant sites of disease progression, such as lungs or intra-parenchymal liver. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as an increase in peritoneal cancer index (PCI) score of greater than 4 points from baseline PCI. New ascites requiring repeat (more than 1) therapeutic paracentesis, malignant bowel obstruction, new intraperitoneal nodules or masses concerning for peritoneal metastasis, and decline in performance status not attributable to other medical causes.
Time Frame: From start of treatment to until time of extra-peritoneal progression, an average of 1 year
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible. This outcome measure was not reported with an 80% confidence interval as required by the protocol because only one participant ever experienced extra peritoneal progression and a median could not be calculated.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With Intra-peritoneal Progression Free Survival (iPFS)
Description: iPFS was determined based on identification of only intraperitoneal sites such as new, malignant ascites, peritoneal nodules, or ovarian metastases. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progression is defined as an increase in peritoneal cancer index (PCI) score of greater than 4 points from baseline PCI. New ascites requiring repeat (more than 1) therapeutic paracentesis, malignant bowel obstruction, new intraperitoneal nodules or masses concerning for peritoneal metastasis, and decline in performance status not attributable to other medical causes.
Time Frame: At extra-peritoneal progression, an average of 1 year
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Participants | 1 | 0

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 3
Population: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
Number analyzed (Participants) | 4 | 7
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, 18 months and 8 days; and 25 months and 10 days for the first and second group, respectively.
Description: 4/5 participants are analyzed in the first group because one participant was deemed ineligible.
Arm/Group | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/7
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/7
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily (N=4) | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily (N=7)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Intraperitoneal 20mg & Intravenous 80mg Every 3Weeks & Capecitabine 825mg/m^2 Twice Daily (N=4) | Paclitaxel Intraperitoneal 60mg & Intravenous 80mg Every 3Weeks &Capecitabine 825mg/m^2 Twice Daily (N=7)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (7) | 1 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (11) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, Covid-19 (Infections and infestations) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (6) | 5 (11)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT04034251/Prot_SAP_002.pdf
  • Informed Consent Form: Cohort: Affected Patients (English) Consent (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT04034251/ICF_001.pdf